CLINICAL TRIAL: NCT05597696
Title: Evaluation of Sitting Balance in Lower Limb Amputees: a Case Control Study
Brief Title: Sitting Balance in Lower Limb Amputees
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gökhan Karakaş, Principal Investigator, Hacettepe University
Other Study IDs: GO 22-385
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Amputation; Traumatic Amputation of Lower Extremity
Keywords: Limits of stability; Sitting balance; Standing balance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1) Experimental Group: Transfemoral Amputee: Balance assessment in sitting
- 2) Control Group: Healthy Subjects: Balance assessment in sitting

SUMMARY:
The aim of this study is to compare the sitting and standing postural stability of transfemoral individuals with healthy individuals with similar demographic characteristics.

DETAILED DESCRIPTION:
Postural stability is important for amputees to perform daily life activities and participate in social activities. The aim of this study is to compare the sitting and standing stability of transfemoral individuals with healthy individuals with similar demographic characteristics. A force platform was used to measure the postural stability of individuals. The sitting limits of stability of the participants were recorded in cm. Amputees between the ages of 18-50, using their prosthesis for at least 6 months, and healthy individuals with similar demographic characteristics were included in the study. Congenital amputees, individuals with bilateral lower extremity amputations, and individuals with central or peripheral vestibular disorders were excluded. Our study will reveal the importance of sitting stability limits in the evaluation and treatment of amputees.

ELIGIBILITY:
Inclusion Criteria for amputee:

* Unilateral transfemoral amputation
* Using their prosthesis for at least 6 months

Exclusion Criteria:

* congenital amputee
* Bilateral lower extremity amputation
* Central or peripheral vestibular disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Amputees who applied to our faculty for prosthesis construction and control, and healthy individuals from relatives of the researcher reached by snowball method will constitute the sample of the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Limits of stability | 15 minutes
  Limits of stability test evaluates dynamic balance of participants. Computerized balance system measured limits of stability for forward, backward, right and left side movements in sitting. It calculates the maximum distance a person can lean without losing balance. The unit of measure is centimeters. The higher value is indicated the better balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Department of Physiotherapy and Rehabilitation, Ankara, Samanpazarı, Turkey (Türkiye)